CLINICAL TRIAL: NCT05414981
Title: A Randomized, Blinded, Placebo-Controlled, Dose-Ranging Phase 1b Study of the Safety, Pharmacokinetics, and Antiviral Activity of ABI-H3733 in Subjects With Chronic Hepatitis B Virus Infection
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Antiviral Activity of ABI-H3733 in Subjects With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABI-H3733-102; 2022-000318-32 (EudraCT Number)
Record Dates: First submitted 2022-06-02; First posted 2022-06-10 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Chronic Hepatitis B
Keywords: cHBV; HBV; Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABI-H3733 (Active Comparator)
  Interventions: Drug: ABI-H3733
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABI-H3733 — 25 mg or 100 mg tablets for oral administration
  Arms: ABI-H3733
Drug: Placebo — 25 mg or 100 mg tablets for oral administration
  Arms: Placebo

SUMMARY:
This is a randomized, blinded, placebo-controlled, dose-ranging Phase 1b study of the safety, PK, and antiviral activity of ABI-H3733 in treatment-naïve or off-treatment chronic Hepatitis B virus (cHBV) subjects that are Hepatitis B e antigen (HBeAg) positive or negative. The study will enroll up to 5 sequential cohorts of 10 subjects each, for a total of up to 50 subjects, randomized 8:2 to receive ABI-H3733 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 18.0 and < 35.0 kg/m(2), where BMI = weight (kg)/(height [m])(2) with a minimum body weight of 45 kg.
2. Chronic hepatitis B infection, defined as HBV infection for ≥6 months documented
3. Treatment-naïve or off-antiviral therapy for ≥24 weeks prior to Screening
4. Lack of bridging fibrosis or cirrhosis

Exclusion Criteria:

1. Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis D virus (HDV), acute hepatitis A virus (HAV), or acute hepatitis E virus (HEV)
2. History of liver transplant or evidence of advanced liver disease, cirrhosis, or hepatic decompensation
3. Clinically significant diseases or conditions
4. History of hepatocellular carcinoma
5. Current or prior treatment for cHBV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-07 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with adverse events (AEs), premature treatment discontinuation due to AEs, and abnormal laboratory results | Through end of study, up to 56 days

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABI-H3733 in subjects with cHBV | Through treatment period, up to 28 days
Minimum Plasma Concentration (Cmin) of ABI-H3733 in subjects with cHBV | Through treatment period, up to 28 days
Area Under Plasma Concentration-Time Curve (AUC) of ABI-H3733 in subjects with cHBV | Through treatment period, up to 28 days
Time to Maximum Plasma Concentration (Tmax) of ABI-H3733 in subjects with cHBV | Through treatment period, up to 28 days
Elimination half-life (t1/2) of ABI-H3733 in subjects with cHBV | Through treatment period, up to 28 days
To evaluate the effect of food on Cmax of ABI-H3733 in subjects with cHBV | Through treatment period, up to 28 days
To evaluate the effect of food on AUC of ABI-H3733 in subjects with cHBV | Through treatment period, up to 28 days
To evaluate the effect of food on the proportion of subjects with AEs, premature discontinuation due to AEs and abnormal laboratory results | Through treatment period, up to 28 days
To evaluate the changes in HBV DNA (IU/mL or Log IU/mL) in subjects with cHBV by Quantitative PCR | Through treatment period, up to 28 days

CONTACTS AND LOCATIONS:
Locations (9):
- Bulgaria (3):
  - Diagnostic Consultative Center Aleksandrovska, Sofia, Sofia-Grad
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia
- University of Hong Kong, Hong Kong, Hong Kong
- ICS Arensia Exploratory Medicine Republican Clinical Hospital "Timofei Moșneaga"- Hospital, Chisinau, Moldova
- New Zealand Clinical Research, Grafton, Auckland, New Zealand
- Institute of Infectious Diseases - Hospital ARENSIA Exploratory Medicine Research Clinic National Institute of Infectious Diseases "Matei Bals", Bucharest, Romania
- Singapore (2):
  - Clinical Trials and Research Centre, Singapore General Hospital, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No